CLINICAL TRIAL: NCT05000996
Title: The Gut Microbiota in Metabolic Surgery: A Multi-Ethnic, Multi-Omic, Longitudinal Study
Brief Title: Gut Microbiota in Metabolic Surgery
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Danxia Yu, Associate Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: VUMC_IRB#201652; R01DK126721 (NIH)
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Bariatric Surgery Candidate; Cardiovascular Diseases; Type 2 Diabetes; Dyslipidemias; Hypertension; Morbid Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Dyslipidemias; Hypertension; Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Stool; Blood (plasma, serum, white blood cells, and red blood cells); Tissue (subcutaneous adipose, omentum, skeletal, jejunum, and stomach)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric Surgery — Roux-en-Y gastric bypass (RYGB) and vertical sleeve gastrectomy (VSG)

SUMMARY:
Metabolic surgery is an emerging option to treat obesity-related metabolic diseases (e.g., type 2 diabetes) and prevent cardiovascular disease (CVD). Metabolic surgery can profoundly alter the gut microbiota; meanwhile, gut microbiota may affect surgical outcomes. Longitudinal studies that examined pre- to post-surgery changes in gut microbiota and its relation to cardiometabolic health after surgery are limited. Furthermore, few studies have included African Americans, a population with high rates of cardiometabolic diseases. The investigators aim to fill these research gaps by establishing a longitudinal, observational study of metabolic surgery patients and applying multi-omics to identify stool, blood, and/or tissue microbial features related to post-surgery cardiometabolic outcomes. In the current study, the investigators plan to enroll up to 300 patients who undergo metabolic surgery at Vanderbilt University Medical Center and follow them for up to 10 years after surgery. Fasting blood and stool samples will be collected at pre-surgery and 3-month, 1-year, 2-year, and 3-year post-surgery clinical visits. Tissue samples (e.g., biopsies of the liver and adipose and remnants of the stomach) will be collected during operation. Meanwhile, participants will complete a REDCap survey at baseline and 1-year, 2-year, and 3-year post-surgery. Participants' electronic medical records will be used to obtain additional information and facilitate long-term follow-up. The investigators will evaluate pre- to post-surgery changes in the fecal microbiome and fecal and blood levels of metabolites and proteins and the associations of microbiome, metabolites, and proteins with cardiometabolic improvements after surgery. This study will advance our understanding of the role of gut microbiota in metabolic surgery, which may translate into novel approaches to identify and treat obese patients for better cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Be approved and scheduled for metabolic surgery at the Vanderbilt University Medical Center
* Have a history of type 2 diabetes, hypertension, or dyslipidemia
* Be able and willing to provide personal information and biological samples needed for the study

Exclusion Criteria:

* Prior gastric operations
* A history of coronary artery disease, stroke, heart failure, HIV infection, or untreated viral hepatitis
* Chemotherapy or radiotherapy for cancer within 2 years
* Current inflammatory bowel disease or celiac disease
* Vomiting, constipation, or diarrhea within 7 days or use of antibiotics within 2 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to enroll 300 patients who undergo metabolic surgery at the Vanderbilt University Medical Center and follow them up to 10 years after surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Estimated 10-year risk of atherosclerotic cardiovascular disease | From before surgery to 1 to 3-year after surgery to 10-year after surgery
  The 10-year risk of atherosclerotic cardiovascular disease based on the American College of Cardiology/American Heart Association pooled cohort equations, incorporating age, sex, race, systolic blood pressure, total cholesterol, HDL cholesterol, diabetes status, hypertension status, and smoking

SECONDARY OUTCOMES:
Glycated hemoglobin | From before surgery to 1 to 3-year after surgery to 10-year after surgery
Blood pressure | From before surgery to 1 to 3-year after surgery to 10-year after surgery
Blood cholesterol | From before surgery to 1 to 3-year after surgery to 10-year after surgery
  Total, low-density, and high-density lipoprotein cholesterol
Blood inflammatory proteins | From before surgery to 1 to 3-year after surgery to 10-year after surgery
  high-sensitivity C-reactive protein

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt_University MC, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yu D, Shu XO, Howard EF, Long J, English WJ, Flynn CR. Fecal metagenomics and metabolomics reveal gut microbial changes after bariatric surgery. Surg Obes Relat Dis. 2020 Nov;16(11):1772-1782. doi: 10.1016/j.soard.2020.06.032. Epub 2020 Jun 27. PMID 32747219

DOCUMENTS (1):
  • Informed Consent Form (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT05000996/ICF_001.pdf